CLINICAL TRIAL: NCT05949515
Title: Retrospective Evaluation of SuperSaturated Oxygen (SSO2) Therapy Clinical Utility (RESCU). An Analysis of Clinical Outcomes and Left Ventricular Recovery of STEMI Patients Treated With SSO2 Therapy After Primary Percutaneous Coronary Intervention (PPCI)
Brief Title: Retrospective Evaluation of SuperSaturated Oxygen (SSO2) Therapy Clinical Utility
Acronym: RESCU
Status: Completed | Type: Observational
Sponsor: Cardiovascular Research Foundation, New York (Other)
Responsible Party: Sponsor
Other Study IDs: RESCU
Record Dates: First submitted 2023-06-28; First posted 2023-07-18 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Acute ST Segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Minneapolis Heart Institute
- The Feinstein Institutes for Medical Research
- NCH Baker Downtown Hospital
- OhioHealth Research Institute
- Baptist Health Baptist Hospital
- St. Mary's Medical Center
- Corewell Health William Beaumont University Hospital - Research Institute
- University of Chicago Medicine

SUMMARY:
The purpose of this multicenter study is to assess the impact of SSO2 treatment on clinical outcomes and left ventricular function in patients following acute ST-segment elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
The TherOx® Downstream® System, which is approved for use in the United States (US) by the Food and Drug Administration (FDA) under P170027. The TherOx® Downstream® System consists of three primary components. These include a hardware device called the TherOx Downstream System ("console"), a single-use disposable device called the TherOx Downstream Cartridge ("cartridge") and a 5 French, commercially available qualified SSO2 infusion coronary delivery catheter ("delivery catheter").

This is a multicenter, retrospective case-control study which will collect data from all STEMI patients who received SSO2 treatment at participating centers, along with up to 3 matched control patients who did not receive SSO2 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Data from all patients who received SSO2 treatment and have completed a minimum of 3 months follow up will be collected at each participating center; there are no other exclusion criteria aside from date of treatment.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a multicenter, retrospective case-control study which will collect data from all STEMI patients who received SSO2 treatment at participating centers, along with up to 3 matched control patients who did not receive SSO2 treatment.
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change of Left Ventricular Ejection Fraction | Baseline to 3 months
  Between group comparison
Rate of Cardiovascular related Hospitalizations | Through study completion, an average of 1 year
  Between group comparison

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Baptist Hospital of Miami, Inc and Its Miami Cardiac and Vascular Institute, Miami, Florida
  - NCH Healthcare System, Naples, Florida
  - Oakwood Healthcare, Inc, Dearborn, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Northwell Health, Inc, Great Neck, New York
  - OhioHealth Research Institute, Columbus, Ohio
  - Avita Health, Galion, Ohio
  - St. Mary's Medical Center, Huntington, West Virginia